CLINICAL TRIAL: NCT06912854
Title: Sensory Adapted Dental Environments to Enhance Oral Care for Children With and Without Dental Fear and Anxiety
Acronym: SADE-DFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Leah Stein Duker, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CHLA-24-00096; UH3DE031222 (NIH)
Record Dates: First submitted 2025-03-18; First posted 2025-04-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Dental Fear and Anxiety
Keywords: sensory adapted dental environment; video-based modeling; dental care; dental anxiety; dental fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four study conditions for their first dental cleaning and then be randomly assigned to one of the three remaining study conditions for their second dental cleaning. We will randomize to treatment order and use counterbalancing, statistically adjust for order of cleaning (i.e., first vs. second cleaning), and covary for any significant interactions between order of cleaning and treatment condition.
Who Masked: Outcomes Assessor
Masking Description: Due to the practicalities of this study and the need to (or not to) modify dental environments and/or provide modeling videos for each participant, blinding of treatment condition for patients or dentists is not applicable. However, for EDA recordings, research team members analyzing/coding data will be masked to condition (SADE, VBM, VBM-SADE, RDE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Regular Dental Environment (RDE) (No Intervention): Participants randomized to a RDE will have their dental cleaning administered in a traditional manner (oral examination, prophylaxis, fluoride application) using tell-show-do and basic behavior guidance techniques including positive reinforcement.
- Video-based Modeling (VBM) (Experimental): Participants randomized to VBM will view a 5-minute video on an iPad that depicts a dental cleaning (oral examination, prophylaxis, and fluoride varnish application) being performed on a sex and age-matched (6-9 yrs v.s 10-12 yrs) cooperative child. This video will feature the model beginning in the waiting room, undertaking a successful cleaning in the absence of any signs of anxiety, choosing a small toy from the dental clinic treasure box, and receiving parental and dentist praise for good behavior.
  Interventions: Other: Video-based Modeling
- Sensory Adapted Dental Environment (SADE) (Experimental): Participants randomized to the SADE will receive their dental cleaning in a environment in which modifications have been made to visual, auditory, and deep pressure (tactile) stimuli to minimize sensory-related discomforts and maximize relaxation. Visual adaptations include: all direct overhead fluorescent lighting and dental overhead lamp will be turned off; black-out curtains will cover the windows; and application of adapted lighting, which will include slow moving visual color effects (Snoezelen) and the dentist wearing a surgical dental headlamp to direct light into the child's mouth, not eyes. Auditory stimuli will include calming rhythmic music projected via portable speakers. Tactile deep pressure stimuli will be provided via a commercially available weighted blanket placed on the child to provide deep "hugging" pressure, which produces a calming effect.
  Interventions: Other: Sensory Adapted Dental Environment
- Video-based Modeling + Sensory Adapted Dental Environment (VBM-SADE) (Experimental): Participants randomized to VBM-SADE will view a modeling video prior to their dental cleaning (see Video-based Modeling description) and experience their dental cleaning in a sensory adapted dental environment (see Sensory Adapted Dental Environment description); the pre-cleaning modeling video will portray the same procedural content as in the VBM-only condition, but with the SADE modifications made to the room in which the child actor receives his/her cleaning.
  Interventions: Other: Sensory Adapted Dental Environment; Other: Video-based Modeling

INTERVENTIONS:
Other: Sensory Adapted Dental Environment — The SADE condition consists of physical adaptations (visual, auditory, tactile modifications) to the dental environment meant to create a less anxiety-provoking sensory experience. Direct overhead fluorescent lighting and the regular dental overhead lamp will be turned off and darkening curtains will cover the windows. Adapted lighting will include slow moving visual color effects (Snoezelen) shining on the ceiling in the child's visual field. The dentist will wear a surgical dental headlamp directed into the patient's mouth, reducing bright lights shining in the child's eyes. Auditory stimuli will be calming rhythmic music (Dan Gibson's Exploring Nature) projected via portable speakers. The tactile deep pressure stimulus will be a commercially available weighted blanket (10-15% of the child's weight) placed on the child to provide deep "hugging" pressure, which produces a calming effect.
  Arms: Sensory Adapted Dental Environment (SADE); Video-based Modeling + Sensory Adapted Dental Environment (VBM-SADE)
Other: Video-based Modeling — Participants will watch an approximately 5-minute video depicting a dental cleaning being performed on a sex and age-matched cooperative child, designed to expose the participant to the activities of the dental cleaning and thereby create a less anxiety-provoking dental experience.
  Arms: Video-based Modeling (VBM); Video-based Modeling + Sensory Adapted Dental Environment (VBM-SADE)

SUMMARY:
This study is a randomized clinical trial investigating the effectiveness of a Sensory Adapted Dental Environment (SADE) alone and together with a video-based modeling (VBM) component (VBM-SADE), compared to a regular dental environment (RDE) and/or VBM alone, to reduce anxiety, distress behavior, pain, and sensory discomfort during a dental cleaning in children with and without dental fear and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 6 through 12 years, of any race/ethnicity;
* English- or Spanish-speaking child and parent;
* Have experienced at least one prior dental cleaning;
* If recruited from the emergency department, Emergency Severity Index (ESI) must be level V or IV (to ensure that greater severity PED patients not be recruited).

Exclusion Criteria:

* Dental cleaning within the previous 4 months (i.e., not in need of cleaning);
* Plan to move out of the area within 6 months;
* Intellectual or developmental disability (e.g. autism; highly co-morbid with sensory processing difficulties);
* Disability that would interfere with oral care (e.g. cleft lip/palate, cerebral palsy, genetic/endocrine/metabolic dysfunction) or medical condition that would place the child at increased risk during the study (e.g., uncontrollable seizures);
* Daily use of anti-cholinergic drugs (i.e., interferes with EDA recordings);
* Presence of orthodontia (braces) or with a plan to get braces in the upcoming 6 months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 312 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Electrodermal Activity (EDA; Skin Conductance Level [SCL]) | Periprocedural
  Electrodermal Activity (EDA; skin conductance level [SCL]) reflects the activation of the sympathetic 'fight or flight' nervous system and is well-documented to increase in stressful or painful situations. A BIOPAC MP160 System will be used to record the child's EDA. The child will relax in dental chair for three minutes in order to obtain a resting baseline EDA measurement, followed by EDA recording for the duration of the dental cleaning.
Electrodermal Activity (EDA; Non-specific Skin Conductance Responses [NS-SCR]) | Periprocedural
  Electrodermal Activity (EDA; frequency of non-specific skin conductance responses [NS-SCR]) reflects the activation of the sympathetic 'fight or flight' nervous system and is well-documented to increase in stressful or painful situations. A BIOPAC MP160 System will be used to record the child's EDA. The child will relax in dental chair for three minutes in order to obtain a resting baseline EDA measurement, followed by EDA recording for the duration of the dental cleaning.
Frequency of Distress Behaviors | Periprocedural
  Frequency of distress behaviors will be scored from video-recordings of the dental cleanings. A trained research team member will assess the count of mouth movements, head movements, and verbal distress behaviors (whimper/cry/scream).
Duration of Distress Behaviors | Periprocedural
  Duration of distress behaviors will be scored from video-recordings of the dental cleanings. A trained research team member will assess the duration of verbal distress behaviors (whimper/cry/scream).

SECONDARY OUTCOMES:
Frankl Scale | Collected immediately after each dental cleaning
  The Frankl Scale is a reliable and valid dentist-report measure categorizing the child's (patient's) behavior during the dental encounter into 4 categories/levels of collaboration starting from rating 1 (definitely negative) to rating 4 (definitely positive). Higher scores indicate higher levels of cooperation during dental treatment.
Anxiety and Cooperation Scale | Collected immediately after each dental cleaning
  The Anxiety and Cooperation Scale is a reliable and valid dentist-report measure rating the child's (patient's) level of anxiety and cooperation using a 6-point numeric scale. Higher scores indicate higher levels of anxiety and lower levels of cooperation.
Wong Baker Faces Pain Scale | Collected immediately after each dental cleaning
  The Wong Baker Faces Pain Scale is a valid tool comprised of six faces to assess perception and intensity of pain. This is a self-report measure with scores ranging from 0-10. Higher scores indicate higher levels of pain.
Dental Sensory Sensitivity Scale | Collected immediately after each dental cleaning
  The Dental Sensory Sensitivity Scale is a self-report measure of the presence and magnitude of discomfort with different sensory stimuli in the environment with scores ranging from 0-12. Children rate 6 items on a 0-2 scale of how much the stimuli bothered them (not at all [0]; a little [1]; a lot [2]) after a dental encounter. Higher scores indicate greater sensory discomfort during routine dental treatment.
Subjective Thoroughness of Cleaning Scale | Collected immediately after each dental cleaning
  The Subjective Thoroughness of Cleaning Scale describes the efficacy of the dental encounter, as perceived by the dentist, and documents the presence/absence of behavioral issues and whether or not they impeded care. Scores range from 0-13 with higher scores indicating a more thorough cleaning.
Client Satisfaction Questionnaire | Collected immediately after each dental cleaning
  The Client Satisfaction Questionnaire is a reliable and valid self-report measure used to assess client/patient perception of satisfaction with services and clinical care. Items are rated on a 4-point Likert scale with varying response options (e.g., 1 = "poor" to 4 = "fair"; 1 = "quite dissatisfied" to 4 = "very satisfied"). Scores range from 8-32 with higher scores indicating greater satisfaction.
Child Intervention Experience Form | Collected immediately after each dental cleaning
  The Child Intervention Experience Form is a self-report measure of how much the child liked the intervention-related adaptations to their dental encounter. Scores range from 1-45 with higher scores indicating a more positive experience.
Caregiver Intervention Experience Form | Collected immediately after each dental cleaning
  The Caregiver Intervention Experience Form is a self-report a measure of how much the caregiver liked the intervention-related adaptations to the dental encounter for their child. Scores range from 1-75 with higher scores indicating a more positive experience.
Dentist Intervention Experience Form | Collected immediately after each dental cleaning
  The Dentist Intervention Experience Form is a measure of how much the dentist liked the intervention-related adaptations to the dental encounter, both for their patient and themselves. Scores range from 10-51 with higher scores indicating a more positive experience.
State-Trait Anxiety Inventory - Short Form | Collected immediately after each dental cleaning
  The State Trait Anxiety Inventory Short Form is a commonly used reliable and valid self-report measure to assess an individual's state and trait anxiety. Items are scored on a 4-point Likert scale with scores ranging from 20 - 80. Higher scores indicate higher levels of state and trait anxiety.
Stress Appraisal Measure | Collected immediately after each dental cleaning
  The Stress Appraisal Measure is a comprehensive tool to measure an individual's appraisal of stress. Items are scored on a 5-point Likert scale with scores ranging from 28 - 140. Higher scores indicate higher stress.
Semi-Structured Interview of Dentists | Through study completion, an average of 1 year
  The Semi-structured Exit Interview of Dentists is a tool to obtain qualitative information about their participation and perception of the study interventions.
Children's Fear Survey Schedule - Dental Subscale | Collected prior to participant's first dental cleaning
  The Children's Fear Survey Schedule-Dental Subscale is a reliable and valid self- or caregiver-report measure to assess dental fear and anxiety in children. Items are scored on a 5-point Likert scale with scores ranging from 12-75. Higher scores indicate greater dental fear and anxiety. A score of less than 32 indicates non-clinical range, scores between 32-38 indicate borderline range, and scores greater than or equal to 39 indicial clinical range of dental fear and anxiety.
Short Sensory Profile | Collected prior to participant's first dental cleaning
  The Short Sensory Profile is a reliable and valid caregiver-report measure to collect information about how children respond to sensory input in daily life activities. Scores at or above 1 standard deviation below the mean indicate typical sensory symptoms. Score at or above the point 2 SD below the mean, but lower than 1 SD below the mean indicate a possible difference in sensory symptoms. Scores below the point 2 SD below the mean indicate a definite difference in sensory symptoms.

OTHER OUTCOMES:
Cleaning Duration | Periprocedural
  Overall duration of time required to complete dental cleaning (oral examination, prophylaxis, fluoride application); scored from video-recording.
Added Procedural Costs | Periprocedural
  Sum of costs due to required additional personnel, protective stabilization, pharmacologic intervention (sedation or general anesthesia).

CONTACTS AND LOCATIONS:
Overall Officials: Leah Stein Duker, PhD, OTR/L, Principal Investigator — University of Southern California
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No